CLINICAL TRIAL: NCT01200407
Title: AN OPEN LABEL, NON-INTERVENTIONAL STUDY OF THE SAFETY, TOLERABILITY, AND EFFICACY OF AMLODIPINE AND OLMESARTAN MEDOXOMIL (NORMETECTM) IN FILIPINO PATIENTS WITH HYPERTENSION: A POST MARKETING SURVEILLANCE STUDY
Brief Title: Amlodipine And Olmesartan Medoxomil In Hypertensive Filipino Patients
Status: Terminated | Type: Observational
Why Stopped: The requirement for Post Marketing Surveillance was lifted by the Philippine FDA
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1581001
Record Dates: First submitted 2010-08-25; First posted 2010-09-13 (Estimated); Results first posted 2021-08-17 (Actual); Last update posted 2021-08-17 (Actual); Status verified 2021-07

CONDITIONS: Hypertension
Keywords: Hypertension; fixed drug combination; Filipinos; Amlodipine; Olmesartan medoxomil; uncontrolled hypertension; difficult to treat hypertension
MeSH Terms: conditions — Hypertension | interventions — Amlodipine; Olmesartan Medoxomil

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Filipino Hypertensive patients: Male and Female, 18 to 65 year old Filipino hypertensive patients prescribed by their doctors with Normetec
  Interventions: Drug: Amlodipine + Olmesartan medoxomil

INTERVENTIONS:
Drug: Amlodipine + Olmesartan medoxomil — start dose is 5/20 mg, which can then be uptitrated to 5/40 mg up to 10/40 mg if BP goal is not reached during the 4 week follow-up

SUMMARY:
The purpose of this study is to determine the safety, tolerability and efficacy of Amlodipine and Olmesartan medoxomil among Hypertensive Filipino patients.

ELIGIBILITY:
Inclusion Criteria:

* Filipino hypertensive subjects ages 18-65 years old whether naive or currently taking any other anti-hypertensive or those on monotherapy using CCBs or ARBs whom they want to shift on a fixed dose combination drug

Exclusion Criteria:

* Patients with contraindications to any of the component of the fixed drug (amlodipine or olmesartan medoxomil) or with malignant or secondary hypertension

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Filipino Hypertensive patients ages 18-65 years old
Sampling Method: Non-Probability Sample
Enrollment: 615 (Actual)
Dates: Start 2010-06-09 (Actual); Primary Completion 2014-01-04 (Actual); Study Completion 2014-01-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (52):
- Philippines (52):
  - Lorma Medical Center, San Fernando City, LA Union
  - Holy Child Hospital, Taclobo, Dumaguete City, Negros Oriental
  - Private Clinic, Albay
  - Private Clinic, Angono
  - Pines City Doctors Hospital, Baguio City
  - Private Clinic, Baguio City
  - Private Clinic, Bulacan
  - Private Clinic, Calamba
  - Private Clinic, Cavite
  - Private Clinic, Cebu
  - Private Clinic, Cebu City
  - Private Clinic, City of Muntinlupa
  - Private Clinic, City of Taguig
  - Private Clinic, Dagupan
  - Private Clinic, Davao City
  - Private Clinic, Eastwood
  - Private Clinic, Iloilo City
  - Private Clinic, Isabela
  - Private Clinic, Kalibo Aklan
  - Private Clinic, Laguna
  - Private Clinic, Laoag
  - Jesus Nazarene General Hospital, Lingayen, Pangasinan
  - Private Clinic, Makati
  - Makati Medical Center, Makati City
  - Private Clinic, Makati City
  - Private Clinic, Mandaluyong
  - Healthway Medical Clinic, Manila
  - Isaac and Catalina Medical Center, Manila
  - Metropolitan Medical Center Institutional Review Board, Manila
  - Metropolitan Medical Center, Manila
  - Private Clinic, Manila
  - The Medical City, Manila
  - Private Clinic, Marikina City
  - Private Clinic, Metro Manila
  - Private Clinic, Nueva Vizcaya
  - Private Clinic, Olongapo City
  - Private Clinic, Pampanga
  - Private Clinic, Paranaque City
  - Private Clinic, Pasay
  - Private cCinic, Pasig
  - Private Clinic, Pasig
  - Dr. Agnes Vargas, Pasig Ciy
  - Private Clinic, Puerto Princesa City
  - Armed Forces of the Philippines Medical Center, Quezon City
  - Private Clinic, Quezon City
  - Angono Medics, Rizal
  - Private Clinic, San Juan City
  - Private Clinic, Tacloban City
  - Private Clinic, Tarlac City
  - Private Clinic, Tugegarao
  - Priavte Clinic, Tuguegarao City
  - Private Clinic, Tuguegarao City

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B1581001&StudyName=Amlodipine%20And%20Olmesartan%20Medoxomil%20In%20Hypertensive%20Filipino%20Patients

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The diagnostic criteria of hypertension (defined by Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure [JNC VII] as systolic blood pressure [BP] >=140 mmHg and diastolic BP >=90 mmHg) and the dosage of study medication were consistent with the investigator's routine clinical setting.
Groups:
- Normetec: Amlodipine/olmesartan medoxomil(Normetec) was prescribed and administered at the recommended starting dose of 5/20 milligrams (mg) once daily according to approved product information in the Philippines.
Period: Overall Study
Arm/Group | Normetec
Started | 615
Completed | 533
Not Completed | 82
Not completed — Lost to Follow-up | 56
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 4
Not completed — Other | 19

BASELINE CHARACTERISTICS:
Population: The full analysis set included all subjects who received at atleast 1 dose of amlodipine and olmesartan medoxomil.
Arm/Group | Normetec
Number analyzed (Participants) | 613
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.7 (11.0)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 334
  Male | 277
  Unspecified | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 610
  Unspecified | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last study drug administration (Week 12) that were absent before treatment or that worsened relative to pre-treatment state. AEs included both SAEs and non-SAEs.
Time Frame: Baseline up to 28 days after last study drug administration (Week 12)
Population: The safety analysis population included all participants who received at least 1 dose of study medication during the observation period.
Measure: Number; unit: participants
Arm/Group | Normetec
Number analyzed (Participants) | 613
participants
  Number of Participants with AEs | 6
  Number of Participants with SAEs | 0

2. Primary Outcome: Change From Baseline in SBP and DBP at Week 12 With Last Observation Carried Forward (LOCF)
Time Frame: Baseline, Week 12
Population: The full analysis population included all participants who received at least 1 dose of study medication during the observation period; number analyzed=number of participants with observed value in category. LOCF method was used to impute missing values.
Measure: Mean (Standard Deviation); unit: millimeters of mercury (mmHg)
Arm/Group | Normetec
Number analyzed (Participants) | 613
millimeters of mercury (mmHg)
  Baseline: SBP: number analyzed (Participants) | 575
  Baseline: SBP | 161.6 (16.04)
  Baseline: DBP: number analyzed (Participants) | 575
  Baseline: DBP | 98.9 (9.33)
  Change at Week 12: SBP LOCF: number analyzed (Participants) | 574
  Change at Week 12: SBP LOCF | -35.8 (16.74)
  Change at Week12: DBP LOCF: number analyzed (Participants) | 574
  Change at Week12: DBP LOCF | -19.4 (10.39)
Statistical Analysis 1: Comparison: Normetec; SBP with LOCF (Week 12); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -35.8, 95% CI 2-sided [-37.2 to -34.4]
Statistical Analysis 2: Comparison: Normetec; DBP with LOCF (Week 12); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -19.4, 95% CI 2-sided [-20.3 to -18.6]

3. Secondary Outcome: Change From Baseline in Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP) at Weeks 4, 8 and 12 Without (w/o) LOCF
Time Frame: Baseline, Week 4, Week 8, Week 12
Population: The full analysis population included all participants who received at least 1 dose of study medication during the observation period; number analyzed=number of participants with observed value in category.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Normetec
Number analyzed (Participants) | 613
mmHg
  Change at Week 4: SBP w/o LOCF: number analyzed (Participants) | 551
  Change at Week 4: SBP w/o LOCF | -24.7 (16.33)
  Change at Week 4: DBP w/o LOCF: number analyzed (Participants) | 551
  Change at Week 4: DBP w/o LOCF | -13.2 (9.46)
  Change and Week 8: SBP w/o LOCF: number analyzed (Participants) | 506
  Change and Week 8: SBP w/o LOCF | -33.0 (16.36)
  Change and Week 8: DBP w/o LOCF: number analyzed (Participants) | 506
  Change and Week 8: DBP w/o LOCF | -17.6 (9.99)
  Change and Week 12: SBP w/o LOCF: number analyzed (Participants) | 423
  Change and Week 12: SBP w/o LOCF | -36.3 (16.64)
  Change and Week 12: DBP w/o LOCF: number analyzed (Participants) | 423
  Change and Week 12: DBP w/o LOCF | -19.9 (9.99)
Statistical Analysis 1: Comparison: Normetec; SBP w/o LOCF (Week 4); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -24.7, 95% CI 2-sided [-26.1 to -23.4]
Statistical Analysis 2: Comparison: Normetec; SBP w/o LOCF (Week 8); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -33.0, 95% CI 2-sided [-34.4 to -31.6]
Statistical Analysis 3: Comparison: Normetec; SBP w/o LOCF (Week 12); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -36.3, 95% CI 2-sided [-37.9 to -34.7]
Statistical Analysis 4: Comparison: Normetec; DBP w/o LOCF (Week 4); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -13.2, 95% CI 2-sided [-14.0 to -12.4]
Statistical Analysis 5: Comparison: Normetec; DBP w/o LOCF (Week 8); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -17.6, 95% CI 2-sided [-18.4 to -16.7]
Statistical Analysis 6: Comparison: Normetec; DBP w/o LOCF (Week 12); Test type: Superiority or Other; p = 0.000, t-test, 2 sided; Mean Difference (Net) = -19.9, 95% CI 2-sided [-20.8 to -18.9]

4. Secondary Outcome: Percentage of Participants Achieving JNC VII Recommended Blood Pressure Goal at Week 12 With LOCF
Description: Based on JNC VII, the ultimate public health goal of antihypertensive therapy is to reduce cardiovascular and renal morbidity and mortality. The JNC VII recommended BP goal is <140/90 mmHg and <130/80 mmHg for participants with diabetes.
Time Frame: Baseline, Week 12
Population: The full analysis population included all participants who received at least 1 dose of study medication during the observation period.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Normetec
Number analyzed (Participants) | 613
percentage of participants | 70.5 [66.9 to 74.1]

ADVERSE EVENTS:
Time Frame: Baseline up to 28 days after last study drug administration (Week 12)
Arm/Group | Normetec
Serious Adverse Events (participants affected / at risk) | 0/613
Other Adverse Events (participants affected / at risk) | 6/613
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Normetec (N=613)
Vertigo positional (Ear and labyrinth disorders) | 1
Chest Pain (General disorders) | 1
Oedema peripheral (General disorders) | 1
Drug hypersensitivity (Immune system disorders) | 1
Dizziness (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1

LIMITATIONS AND CAVEATS:
This was an observational, non-interventional study which evaluated Filipino patients with hypertension at the outpatient clinic, and as such, study medication was prescribed at the discretion of the attending physician.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single enter publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.